CLINICAL TRIAL: NCT01617031
Title: Biological Efficacy of Twice Daily Aspirin in Type 2 Diabetic Patients With Coronary Artery Disease
Brief Title: Aspirin Twice Daily in Diabetic Patients With Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Dr Jean-Guillaume DILLINGER, Medical Doctor in the Department of Cardiology, Principal Investigator, Assistance Publique - Hôpitaux de Paris
Other Study IDs: LRB-10-023
Record Dates: First submitted 2012-05-25; First posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes Mellitus
Keywords: aspirin; diabetes mellitus; coronary artery disease
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetic patients with coronary artery disease: Type 2 diabetic patients with previous coronary artery disease. All patients are routinely treated with aspirin in secondary prevention of cardiovascular disease. Coronary artery disease is defined as a previous coronary angiography with at least 1 coronary artery stenosis >50%. Type 2 diabetes is defined as patients with diabetes discovered after 30 years old and insulin was not the first treatment except in case of acute coronary syndrome.

SUMMARY:
The aim of the study is to evaluate platelet function variations according to the delay since last aspirin intake (12 vs 24 hours)in a population of diabetic patients with previous Coronary Artery Disease.

DETAILED DESCRIPTION:
We have previously demonstrated that there was a time-dependant efficacy of aspirin on platelet function. In this study, we investigate platelet function (fundamental research) according to the delay since last aspirin intake (12 vs 24 hours)in a population of diabetic patients with previous Coronary Artery Disease routinely treated with aspirin. In order to eliminate any variation linked to a cumulative dose effect of aspirn, platelet function is assessed 24 hours after a single 150 mg aspirin intake or 12 hours after a 75 mg aspirin intake given twice per day (corresponding to the same total dose of 150 mg /day). Light transmission aggregometry triggered by arachidonic acid 0.5mg/mL (LTA-AA) is the main endpoint of the study (intensity and velocity of agregation following exposure to arachidonic acid 0.5 mg/ml).

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* documented coronary artery disease
* treatment with aspirin for at least 7 days before randomization
* one of the following additional criteria defined from our previous study9: current smoking, hs-CRP > 4mg/L, fibrinogen > 4g/L and/or platelet count > 270 103/mm3

Exclusion Criteria:

* oral anticoagulants, heparin, thrombolytic agents, non-steroidal anti-inflammatory drugs, prasugrel
* family or personal history of bleeding or thrombophilic disorders
* platelet count > 600x103/mm3 or < 150x103/mm3
* hematocrit > 50% or < 25%
* creatinine clearance < 30mL/min
* low compliance before enrollment
* cancer considered not in remission or those having undergone major surgery within the month prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive stable DM patients presenting to the Department of Cardiology, Lariboisiere Hospital. Patients are eligible if they have DM and documented CAD and are treated for at least 7 days with a non-enteric-coated aspirin.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Intensity of platelet agregation following exposure to 0.5 mg/ml arachidonic acid | 10 days
  Flow cytometry study of the intensity of platelet agregation following exposure of Platelet reach plasma to 0.5 mg/ml arachidonic acid

SECONDARY OUTCOMES:
Closure time after exposure of total blood to Collagen-epinephrine | 10 days
  Closure time after exposure of total blood to Collagen-epinephrine using Platelet Function Analyzer-100 (PFA-100) with collagen-epinephrine (EPI) cartridge.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Henry, MD-PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of Cardiology-Lariboisiere Hospital-Assistance Publique-Hôpitaux de Paris, Paris, France